CLINICAL TRIAL: NCT06764758
Title: Short-Term Clinical Comparison of Anxiety Levels With Salivary Cortisol Levels in Patients Undergoing Endodontic and Restorative Treatment
Brief Title: Anxiety Levels of Patients Subjected to Endodontic and Restorative Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: D-KA23/28
Record Dates: First submitted 2025-01-03; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Dental Anxiety
Keywords: dental anxiety; salivary cortisol; dental anxiety scale
MeSH Terms: interventions — Endodontics; Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endodontic treatment (Active Comparator): gutta-percha (Sure Dent Corporation; Gyeonggi-do, Korea)
  Interventions: Procedure: Endodontic treatment
- Restorative treatment (Active Comparator): Composite resin restorative material (3M Espe Filtek; Lake County, Minnesota, USA)
  Interventions: Procedure: Restorative treatment

INTERVENTIONS:
Procedure: Endodontic treatment — Root-canal therapy applied in asymptomatic teeth with deep carious lesion required endodontic treatment.
  Arms: Endodontic treatment
Procedure: Restorative treatment — Composite resin restoration applied in teeth previously applied endodontic treatment.
  Arms: Restorative treatment

SUMMARY:
This study aimed to compare the stress levels induced in patients at the beginning and at the end of endodontic and restorative treatments and access relationship between dental anxiety levels and cortisol levels.

For this study, 44 patients requiring endodontic and restorative treatment on a maxillary premolar tooth were selected. Patients were requested to fill out the Corah Dental Anxiety Scale (CDAS) questionnaire prior to and following each treatment procedure. Saliva samples were then collected using the roll cotton method. The saliva was analysed by using the Liquid Chromatography-Mass Spectrometry/Mass Spectrometry (LC-MS/MS) method. Intragroup comparisons of CDAS and cortisol levels were conducted using the Wilcoxon Signed Rank Test. Intergroup comparisons were performed employing the Mann-Whitney U Test. The magnitude of the association between continuous variables was investigated by calculating Spearman's rank-order correlation coefficients along with corresponding significance levels (p< 0.05).

DETAILED DESCRIPTION:
Anxiety is a psychological state defined as significant worry, fear, and tension in response to perceived threats, dangers, or uncertainties. A key long-term consequence of stress exposure is an increased release of cortisol, a hormone regulated by the activation of the hypothalamic-pituitary-adrenal (HPA) axis and the adrenal glands. Cortisol is integral to the body's stress response, with its levels increasing notably during episodes of anxiety, thereby triggering physiological changes.

Dental anxiety, specifically, refers to an intense fear and apprehension associated with dental treatments. This type of anxiety may be associated with several factors, such as negative dental experience, the nature of dental procedures, or individual perception of treatment. Moreover, demographic factors like socioeconomic status, sex, education, and age can impact the development of dental anxiety. Also, childhood experiences of traumatic dental treatments are another critical factor, often resulting in negative attitudes toward dental care.

Research shows that dental anxiety tends to peak during procedures involving injections, though other treatments like dental restorations, endodontic treatment, and tooth extractions are also major sources of distress. Various approaches are utilized to assess dental anxiety, including measuring cortisol levels, administering self-report questionnaires, and using pain rating scales. Commonly applied tools include the Spielberger State-Trait Anxiety Inventory (STAI), Corah's Dental Anxiety Scale (CDAS), Dental Fear Survey (DFS), and the Modified Dental Anxiety Scale (MDAS).

The null hypothesis proposes that endodontic and restorative procedures evoke similar anxiety levels in patients, with no significant association detected between salivary cortisol levels and CDAS measurements.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years old
* Participants who are classified as ASA I according to the American Society of Anaesthesiologists (ASA) physical status classification system.
* Patients who require root canal treatment and will have composite restoration afterwards.

Exclusion Criteria:

* Patients with communication and cooperation problems.
* Patients who take medication regularly.
* Conditions such as Sjögren's syndrome or xerostomia, which affect salivary flow.
* Pregnancy.
* Patients with systemic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Corah's Dental Anxiety Scale | Day 1 and day 7
  The general anxiety level associated with dental procedures was assessed through the Corah Dental Anxiety Scale (CDAS), which includes of four questions designed to evaluate the patient's dental anxiety level. The results were evaluated using a scoring system ranging from 4 (no anxiety) to 20 (high anxiety).

SECONDARY OUTCOMES:
Salivary Cortisol Levels | Day 1 and day 7
  In evaluating the patients' stress levels through experimental and chemical tests, the method of measuring cortisol levels from salivary samples was preferred. The results were evaluated using a scoring system ranging from 1.4 (low salivary cortisol level) -10.1(high salivary cortisol level) ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Gulsahi, DDS., PhD, Study Chair — Baskent University Faculty of Dentistry
Locations (1):
- Baskent University Faculty of Dentistry, Ankara, Turkey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data will be made available by contacting the first author
Supporting Information: Study Protocol
Time Frame: Data will be available after 6 months after article publication
Access Criteria: for research purposes by contacting the first author via e-mail